CLINICAL TRIAL: NCT03478839
Title: A Natural History Study of Patients With Generalized Arterial Calcification of Infancy (GACI) or Autosomal Recessive Hypophosphatemic Rickets Type 2 (ARHR2)
Brief Title: Study of People With Generalized Arterial Calcification of Infancy (GACI) or Autosomal Recessive Hypophosphatemic Rickets Type 2 (ARHR2)
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 180064; 18-HG-0064
Record Dates: First submitted 2018-03-14; First posted 2018-03-27 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-07-07

CONDITIONS: Generalized Arterial Calcification of Infancy; Autosomal Recessive Hypophosphatemic Rickets Type2
Keywords: Generalized Arterial Calcification of Infancy; Autosomal Recessive Hypophosphatemic Rickets; Pseudoxanthoma Elasticum; Idiopathic Infantile Arterial Calcification; Natural History
MeSH Terms: conditions — Arterial calcification of infancy; Hypophosphatemic Rickets, Autosomal Recessive, 1; Pseudoxanthoma Elasticum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CRF completion: Individuals with a diagnosis of GACI or ARHR2 with sufficient chart data to be included in the study will be eligible for enrollment, as well as all their siblings and parents.

SUMMARY:
Background:

Generalized Arterial Calcification of Infancy (GACI) is a very rare disorder. It can be fatal before birth or by age 6 months. Anumber of people with GACI survive into adulthood. Those adults suffer from side effects of the disease, including rickets. It is unknown how common the disease Autosomal Recessive Hypophosphatemic Rickets Type 2 (ARHR2) is. It also has side effects. GACI and ARHR2 are usually caused by the mutations in the same gene. There are no approved treatments for the two diseases. Researchers want to study people with these diseases and their family members. This may help understand these rare and unique diseases better. The data could lead to new treatments for GACI and ARHR2.

Objectives:

To better understand the progression of GACI and ARHR2 and how genes might play a role in them.

Eligibility:

People with GACI or ARHR2, both living and deceased, and their parents and siblings.

Design:

Participants will allow researchers to access their medical records. They will give this consent by mail, email, or fax.

Data will be taken from the records. Participants names will not be used. Instead, they will be identified by a code.

Participants may give a blood sample.

If a participant withdraws from the study, their data and samples will be destroyed. However, the coded clinical data in the official medical record and data in databases will NOT be destroyed.

...

DETAILED DESCRIPTION:
This is a natural history study of patients with Generalized Arterial Calcification of Infancy (GACI) or Autosomal Recessive Hypophosphatemic Rickets Type 2 (ARHR2).

GACI is an ultra-rare disorder with an estimated birth prevalence of around 1 in 200,000. GACI is characterized by extensive arterial calcifications, arterial stenosis, myointimal proliferation and periarticular calcifications. Individuals with GACI also experience calcification in other body areas, such as joints and parenchymal organs.

GACI is generally fatal before birth or within the first six months after birth. The cause of death is frequently myocardial infarction or stroke, and hypertension and congestive heart failure are common in fetuses and infants with GACI. The first six months of life are considered a critical period for GACI patients, and approximately 85% of infants with GACI do not survive beyond this period (Moran 1975). However, the mortality rate decreases substantially among patients who do survive beyond the critical period. Reports exist of patients with GACI who survived into adulthood, but the frequency of this occurrence is unknown, and adult patients suffer from a number of sequelae such as cognitive impairment related to stroke. ARHR2 is characterized by short stature, dental caries, and bone deformities, and biochemically by hypophosphatemia, hyperphosphaturia and elevated plasma alkaline phosphatase. The disease frequency is unknown.

GACI and ARHR2 are most commonly due to mutations of ENPP1 (ectonucleotide pyrophosphatase/phosphodiesterase 1), or less often from mutations in ABCC6 (adenosine triphosphate binding cassette transporter protein subfamily C member 6). No founder mutations are known, and thus no ethnic predilection is known. Both the GACI and ARHR2 phenotypes are potentially fatal or associated with severe morbidity, with no FDA-approved drugs or proven treatments. Animal data suggest that enzyme replacement therapy with ENPP1-Fc may be effective in preventing morbidity or mortality of GACI and ARHR2.

PXE (pseudoxanthoma elasticum) is an autosomal recessive disorder due to mutations in ABCC6 or, less often, ENPP1. PXE is characterized by ectopic calcification of the skin, eyes, cardiovascular system and gastrointestinal system. This study will not focus on PXE but will collect data on PXE patients, particularly when their presentation suggests elements of the GACI or ARHR2 phenotypes.

The main objective of this study is to collect historical control data for future comparison to data from patients treated with ENPP1-Fc so we can develop ENPP1-Fc as a treatment for GACI or ARHR2. In addition, this study will allow for a better understanding of the disease course to design future treatment trials. The study will utilize data obtained predominantly from chart review. The goal is to enroll 100 participants, which include both living and deceased individuals with GACI or ARHR2, and/or their parents and siblings. Our study will be jointly and collaboratively conducted by the NIH and Inozyme.

ELIGIBILITY:
* INCLUSION & EXCLUSION CRITERIA:

Based upon study purpose, participants enrolled in this protocol must:

1. Have genetic confirmation of one of the following:

   1. GACI due to ENPP1 or ABCC6 mutations
   2. ARHR2 due to ENPP1 mutations
   3. PXE due to ABCC6 or ENPP1 mutations

   AND/OR

   Carry the clinical diagnosis of GACI, ARHR2 or PXE
2. Consent or, if applicable, assent to participate in the study
3. Have sufficient chart information to allow for the completion of at least one of the protocol s objectives.

Ages: 1 Year to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with a diagnosis of GACI or ARHR2 who are males or females with sufficient chart data to be included in the study will be eligible for enrollment, as well as all their male and female siblings and both parents.@@@
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Natural History | ongoing
  The main objective of this study is to determine the natural history of patients with GACI or ARHR2.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos R Ferreira Lopez, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Albright RA, Stabach P, Cao W, Kavanagh D, Mullen I, Braddock AA, Covo MS, Tehan M, Yang G, Cheng Z, Bouchard K, Yu ZX, Thorn S, Wang X, Folta-Stogniew EJ, Negrete A, Sinusas AJ, Shiloach J, Zubal G, Madri JA, De La Cruz EM, Braddock DT. ENPP1-Fc prevents mortality and vascular calcifications in rodent model of generalized arterial calcification of infancy. Nat Commun. 2015 Dec 1;6:10006. doi: 10.1038/ncomms10006. PMID 26624227
- [Background] Ziegler SG, Gahl WA, Ferreira CR. Generalized Arterial Calcification of Infancy. 2014 Nov 13 [updated 2020 Dec 30]. In: Adam MP, Bick S, Mirzaa GM, Pagon RA, Wallace SE, Amemiya A, editors. GeneReviews(R) [Internet]. Seattle (WA): University of Washington, Seattle; 1993-2026. Available from http://www.ncbi.nlm.nih.gov/books/NBK253403/ PMID 25392903
- [Background] Rutsch F, Boyer P, Nitschke Y, Ruf N, Lorenz-Depierieux B, Wittkampf T, Weissen-Plenz G, Fischer RJ, Mughal Z, Gregory JW, Davies JH, Loirat C, Strom TM, Schnabel D, Nurnberg P, Terkeltaub R; GACI Study Group. Hypophosphatemia, hyperphosphaturia, and bisphosphonate treatment are associated with survival beyond infancy in generalized arterial calcification of infancy. Circ Cardiovasc Genet. 2008 Dec;1(2):133-40. doi: 10.1161/CIRCGENETICS.108.797704. PMID 20016754
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2018-HG-0064.html